CLINICAL TRIAL: NCT05123924
Title: Respiratory Functions and Fatigue in Patients With Pediatric-Onset Multiple Sclerosis: A Comparative Cross-sectional Study
Brief Title: Respiratory Functions in Pediatric-Onset Multiple Sclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Yonca Zenginler Yazgan, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: IUC-2021-68
Record Dates: First submitted 2021-11-05; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Pediatric-onset Multiple Sclerosis
Keywords: Pediatric-onset multiple sclerosis; Physiotherapy; Respiratory capacity; Fatigue
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POMS Group: Individuals in the POMS group will be evaluated in terms of respiratory capacity, respiratory muscle strength and fatigue.
  Interventions: Other: Evaluation of respiratory capacity, respiratory muscle strength and fatigue
- Control Group: Individuals in the control group will be evaluated in terms of respiratory capacity, respiratory muscle strength and fatigue.
  Interventions: Other: Evaluation of respiratory capacity, respiratory muscle strength and fatigue

INTERVENTIONS:
Other: Evaluation of respiratory capacity, respiratory muscle strength and fatigue — The demographic information of the participants will be taken with the form prepared for the people in this group. Then, respiratory function with "Minispir Light Spirometer", respiratory muscle strength with "MD Diagnostics RP Check" and fatigue with Pediatric Quality of Life Inventory (PedsQL)-Multidimensional Fatigue Scale will be evaluated. All assessments will be completed on the same day and will not be repeated after a certain period of time.

SUMMARY:
Pediatric-onset multiple sclerosis (POMS) is a chronic, autoimmune and inflammatory disease of the central nervous system that begins before the age of 18 years. POMS patients are affected in terms of physical capacity, cognitive status and fatigue compared with their healthy peers that has been reported. It has been reported that although individuals with MS with low disability levels do not have respiratory complaints, respiratory parameters may be affected. Therefore, it is necessary to evaluate respiratory capacity, respiratory muscle strength and fatigue levels of POMS patients. Evaluations will help prevent future complications by detecting any existing problems early.

DETAILED DESCRIPTION:
People with pediatric onset multiple sclerosis (POMS) may experience sensory, motor, cerebellar and cognitive dysfunctions due to the destruction of the central nervous system. These disorders can cause decrease in physical capacity, increase in cognitive symptoms and fatigue level in patients with POMS. There is no study in the literature examining the relationship between respiratory capacity and respiratory muscle strength with fatigue in POMS patients. The aim of this study is to compare POMS patients and healthy controls in terms of respiratory capacity, respiratory muscle strength and fatigue. All participants's respiratory function will be evaluated with "Minispir Light Spirometer", respiratory muscle strength with "MD Diagnostics RP Check" and fatigue with Pediatric Quality of Life Inventory (PedsQL)-Multidimensional Fatigue Scale. Evaluations will not be repeated after a certain interval.As a result of the comparison of both groups, it will be determined whether POMS patients have difficulties or not.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate
* Being diagnosed with pediatric onset multiple sclerosis
* Being between the ages of 15-22
* EDSS <6

Exclusion Criteria:

* Having another diagnosis in addition to the diagnosis of pediatric-onset multiple sclerosis
* Having a blurred vision problem
* Having had an attack or received corticosteroid treatment 3 months before participating in the study

Ages: 15 Years to 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Thirty patients with POMS who were diagnosed with pediatric-onset multiple sclerosis and met the inclusion criteria will be included in the study. Sample size, Gravesande et al. According to the child form in the PedsQL Multidimensional Fatigue Questionnaire, which they used in their study, according to the total fatigue scores (difference Δ 10.21), in POMS patients (61.57±20.78) and healthy individuals of the same age group (71.78±15.58), with 0.05 margin of error and 80% power. calculated. According to this calculation, it was seen that 25 patients with POMS and 13 healthy individuals who were matched for age and sex (2:1 distribution) should be included in our study.
Sampling Method: Probability Sample
Enrollment: 46 (Estimated)
Dates: Start 2021-10-29 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Evaluation of FEV1/FVC ratio | Baseline
  The Minispir Light Spirometer will be used to assess the respiratory function of the participants. Before starting the spirometric test, how to do the test will be explained. Before starting the test, the participant will be asked to sit with their back straight and put on the nose clip provided. Then the participant will take the disposable bacterial filter mouthpiece between his lips and hold it tightly. The person will be asked to take a few normal breaths followed by as deep a breath as possible and instructed to exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds. If the participant will coughs or cannot breathe deeply enough during the test, the test will terminated and the test will repeated after 20 minutes of rest. The FEV1/FVC ratio with the highest value from three consecutive correctly performed tests will be recorded.

SECONDARY OUTCOMES:
Evaluation of Forced Vital Capacity (FVC) | Baseline
  The Minispir Light Spirometer will be used for FVC evaluation. Before starting the test, it will be explained how to do the test. The participant will be asked to sit with their back straight and put on the nose clip provided. Then the participant will take the disposable bacteria filter mouthpiece between his lips and holds it tightly. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds. If the participant coughs or cannot breathe deeply enough during the test, the test is terminated and the test is repeated after 20 minutes of rest. The highest FVC value from three correctly performed consecutive tests will be recorded.
Evaluation of Forced Expiratory Volume in 1 second (FEV1) | Baseline
  The Minispir Light Spirometer will be used for FEV1 evaluation. Before starting the test, it will be explained how to do the test. The participant will be asked to sit with their back straight and put on the nose clip provided. Then the participant will take the disposable bacteria filter mouthpiece between his lips and holds it tightly. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds. If the participant coughs or cannot breathe deeply enough during the test, the test is terminated and the test is repeated after 20 minutes of rest. The highest FEV1 value from three correctly performed consecutive tests will be recorded.
Evaluation of Peak Expiratory Flow (PEF) | Baseline
  The Minispir Light Spirometer will be used for PEF evaluation. Minispir Light Spirometer will be used for PEF evaluation. Before starting the test, it will be explained how to do the test. The participant will be asked to sit with their back straight and put on the nose clip provided. Then the participant will take the disposable bacteria filter mouthpiece between his lips and holds it tightly. The person will be asked to take a few normal breaths, then take as deep a breath as possible, and then exhale forcefully and quickly without waiting. The test will be terminated by instructing the participant to take a deep breath after exhaling for at least six seconds. If the participant coughs or cannot breathe deeply enough during the test, the test is terminated and the test is repeated after 20 minutes of rest. The highest PEF value from three correctly performed consecutive tests will be recorded.
Evaluation of Respiratory Muscle Strength | Baseline
  Evaluation of respiratory muscle strength will be done with the "MD Diagnostics RP Check" device in accordance with the guidelines of the American Thoracic Society (ATD) and the European Respiratory Society (ASD). The maximum expiratory pressure (MEP) and maximum inspiratory pressure (MIP) of each participant will be measured. Before starting the test, it will be explained how to do the test. During the assessment, the participant will be asked to sit with his back straight and put on the nose clip provided. Then, for the MEP evaluation, the patient will be asked to take a deep breath and blow the whole breath forcefully into the device with a disposable bacteria filter mouthpiece. For the MIP evaluation, the patient will be asked to breathe strongly through the device with a disposable bacteria filter mouthpiece after exhaling the whole breath. Appropriate breaks will be given between assessments. Three correctly performed attempts for MEP and MIP measurements will be recorded.
Pediatric Quality of Life Inventory (PedsQL)-Multidimensional Fatigue Scale | Baseline
  The Pediatric Quality of Life Inventory (PedsQL)-Multidimensional Fatigue Scale is a valid and reliable scale for assessing fatigue in the pediatric population. This 18-item symptom-focused scale evaluates 3 areas of fatigue (general, sleep/rest, and cognitive). Each question is scored on a 5-point Likert system (0=Never, 1=Almost never, 2=Sometimes, 3=Frequently, 4=Always), and high scores indicate higher levels of fatigue. In our study, both the child form and the family form of the scale will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Buket Akıncı, Assoc. Prof., Study Chair — Biruni University; Pelin Vural, MSc., Study Chair — Istanbul University-Cerrahpasa, Graduate Education Institute; Serhat Güler, MD, Study Chair — Istanbul University-Cerrahpasa, Cerrahpasa Faculty of Medicine, Department of Pediatric Neurology
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırköy, Turkey (Türkiye)

REFERENCES:
- [Derived] Vural P, Akinci B, Guler S, Saltik S, Yazgan YZ. Respiratory functions, respiratory muscle strength and fatigue in patients with pediatric-onset multiple sclerosis: a comparative cross-sectional study. Acta Neurol Belg. 2025 Feb;125(1):69-75. doi: 10.1007/s13760-024-02628-4. Epub 2024 Aug 21. PMID 39168946